CLINICAL TRIAL: NCT00003815
Title: A Randomised Study of High Dose Chemotherapy/Radiotherapy and Autologous Bone Marrow Transplantation in Patients With High Grade Malignant Non-Hodgkin's Lymphoma (Kiel Classification) According to Prognostic Groups
Brief Title: Chemotherapy and Radiation Therapy Plus Bone Marrow Transplantation in Treating Patients With Aggressive Non-Hodgkin's Lymphoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Scotland and Newcastle Lymphoma Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000066967; SNLG-NHL-Va; EU-98032
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2001-07

CONDITIONS: Lymphoma
Keywords: stage I adult diffuse mixed cell lymphoma; stage I adult diffuse large cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage I adult lymphoblastic lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Bleomycin; Carmustine; Cyclophosphamide; Cytarabine; Doxorubicin; Etoposide; Melphalan; Prednisolone; Vincristine; Radiotherapy

INTERVENTIONS:
Biological: bleomycin sulfate
Drug: carmustine
Drug: cyclophosphamide
Drug: cytarabine
Drug: doxorubicin hydrochloride
Drug: etoposide
Drug: melphalan
Drug: prednisolone
Drug: vincristine sulfate
Procedure: autologous bone marrow transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage cancer cells. Bone marrow transplantation may allow doctors to give higher doses of chemotherapy drugs and kill more cancer cells.

PURPOSE: Randomized phase III trial to study the effectiveness of chemotherapy and radiation therapy plus bone marrow transplantation in treating patients who have aggressive non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the rate of remission in patients with aggressive non-Hodgkin's lymphoma treated with high-dose chemotherapy and radiotherapy plus autologous bone marrow transplantation.
* Determine the efficacy and toxic effects of this regimen in these patients.

OUTLINE: This is a randomized, placebo-controlled, multicenter study. Patients are stratified according to risk group (good vs intermediate vs poor).

Patients undergo harvest of autologous bone marrow stem cells after priming chemotherapy and before transplantation.

Patients receive induction chemotherapy comprising the CHOP or VAPEC-B regimen. The CHOP regimen consists of vincristine (VCR) IV, cyclophosphamide (CTX) IV, and doxorubicin (DOX) IV on day 1 and oral prednisolone (PRDL) on days 1-5. Treatment repeats every 3 weeks for six courses. The VAPEC-B regimen consists of DOX IV on days 1, 15, 29, 43, 57, and 71; CTX IV on days 1, 29, and 57; VCR IV on days 8, 22, 36, 50, and 64; bleomycin IV on days 8, 36, 64; oral etoposide (VP-16) on days 15-19, 43-47, and 71-75; and oral PRDL daily for 13 weeks.

Patients then may undergo radiotherapy for 2-3 weeks to areas of original bulk or residual disease.

* Good-risk group: Patients are randomized to one of two treatment arms.

  * Arm I: Patients receive no further treatment.
  * Arm II: Patients receive melphalan (L-PAM) before or after total body irradiation (TBI), which is delivered in 3 fractions over 24 hours. After completion of radiotherapy, patients undergo autologous bone marrow transplantation (AuBMT).
* Intermediate- or poor-risk group: Patients are randomized one of three treatment arms.

  * Arm III: Patients receive L-PAM IV on day -2 and AuBMT on day 0.
  * Arm IV: Patients receive treatment as in arm II.
  * Arm V: Patients receive carmustine IV on day -6, VP-16 IV once daily and cytarabine IV twice daily on days -5 to -2, and L-PAM IV on day -1. Radiotherapy to bulk disease begins after completion of chemotherapy. Patients undergo AuBMT on day 0.

Patients are followed monthly for 3 months, every 2 months for 1 year, every 4 months for 2 years, and then every 6 months thereafter.

PROJECTED ACCRUAL: Not specified

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed aggressive non-Hodgkin's lymphoma requiring chemotherapy
* Stage II, III, or IV

  * B cell:

    * Centroblastic
    * Immunoblastic
    * Large cell anaplastic
    * Non-Burkitt lymphoblastic
  * T cell:

    * Pleomorphic medium cell
    * Pleomorphic large cell
    * Immunoblastic
    * Large cell anaplastic
    * Lymphoblastic

      * No Burkitt (L3) subtype
      * No large mediastinal mass OR
* Stage I, II, III, or IV

  * Bulk disease greater than 10 cm
  * Nodal or extranodal site
* No primary localized gut lymphoma
* No CNS involvement

PATIENT CHARACTERISTICS:

Age:

* 15 to 65

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* No concurrent bone marrow dysplastic syndromes

Hepatic:

* Bilirubin no greater than 2.5 times upper limit of normal (ULN)

Renal:

* Creatinine no greater than 2.5 times ULN

Other:

* No other malignancy except skin cancer or stage I cervical cancer
* Not pregnant

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* No prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1994-06

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J. Proctor, MD, FRCP, FRCPath, Study Chair — Newcastle-upon-Tyne Hospitals NHS Trust
Locations (1):
- Newcastle Upon Tyne Hospitals NHS Trust, Newcastle upon Tyne, England, United Kingdom